CLINICAL TRIAL: NCT02170922
Title: Relative Bioavailability of 200 mg Film Coated Tablets of BIBR 1048 MS With or Without Food Compared to 200 mg Solution of BIBR 1048 MS Given as Single Oral Administrations to Healthy Subjects. A 3-way Crossover, Open, Partly Randomized Study.
Brief Title: Bioavailability of BIBR 1048 MS Tablets in Healthy Subjects With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.3
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- Sequence 1 (Experimental): BIBR 1048 MS tablet (fasted) - BIBR 1048 MS solution (fasted) - BIBR 1048 MS tablet after high fat meal
  Interventions: Drug: BIBR 1048 MS tablet; Drug: BIBR 1048 MS solution
- Sequence 2 (Experimental): BIBR 1048 MS solution (fasted) - BIBR 1048 MS tablet (fasted) - BIBR 1048 MS tablet after high fat meal
  Interventions: Drug: BIBR 1048 MS tablet; Drug: BIBR 1048 MS solution

INTERVENTIONS:
Drug: BIBR 1048 MS tablet
Drug: BIBR 1048 MS solution

SUMMARY:
Comparative pharmacokinetics of BIBR 1048 MS solution and tablet with or without food

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 1999-07; Primary Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Maximum plasma concentration (Cmax) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Time from dosing to the maximum concentration (tmax) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug

SECONDARY OUTCOMES:
Change in activated partial thromboplastin time (aPTT) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Change in international normalized ratio (INR) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Terminal half-life (t1/2 ) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Total mean residence time (MRTtot) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Total clearance (CL/f) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug
Volume of distribution (Vz/F) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 48 hours after administration of study drug